CLINICAL TRIAL: NCT05763134
Title: Critical Care Ultrasound Guided Weaning
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Sule Asri, MD, Antalya Training and Research Hospital
Other Study IDs: ultrasound weaning
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-02

CONDITIONS: Weaning Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- weaning failure: Unstable patient without mechanical ventilator support within 48 hours
- weaning success: Stable patient for more than 48 hours without mechanical ventilator support

SUMMARY:
Weaning patients from the ventilator in the intensive care unit is sometimes difficult because of three main interrelated etiologies: impaired lung, heart or diaphragm function. In this context, ultrasonography performed during tests for extubation of patients may enable the diagnosis of cardiac dysfunction, loss of pulmonary aeration, diaphragm dysfunction, and venous congestion, thereby reducing the number of failures in extubation.

The combination of TTE (Trans Thoracic Echocardiography), LUS (Lung Ultrasound), DUS (Diaphragmatic ultrasound) and VEXUS (Venous excess Ultrasound) may enable the identification of the etiology of weaning failure and reduce the number of extubation failures by enabling the development of an appropriate treatment strategy. With this study, it is aimed to contribute to the literature in this sense.

DETAILED DESCRIPTION:
The aim of this study is to reduce the number of extubation failures by defining the etiology of weaning failure and developing appropriate treatment strategies by using intensive care ultrasonography applications in combination (defining cardiac, pulmonary, diaphragmatic and venous congestion).

Most patients can be extubated after the first SBT (spontaneous Breathing Trial). A patient who fails extubation is automatically classified as difficult weaning, and intensive care professionals frequently encounter patients who are difficult to wean from mechanical ventilation.

Before performing a new SBT following a failed SBT, the cause of the failure should be determined and an appropriate treatment strategy developed.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation > 24 hours Eligibility to weaning from mechanical ventilation

Exclusion Criteria:

* Age < 18 years old
* Severe skin lesions or infections that cannot perform ultrasound
* Severe subcutaneous emphysema that cannot perform ultrasound
* Patients with a known neuromuscular disease
* Patients with a duration of mechanical ventilation <24 hours,
* Patients with severe mitral stenosis, severe mitral regurgitation, or prosthetic mitral valve

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The researchers aimed to predict the success and failure of extubation and measure the associated ultrasound indices with the combined ultrasound-guided weaning protocol in all critically ill patients over the age of 18 who remain on mechanical ventilator for more than 24 hours and are thought to be ready for weaning. Evaluations will be made just before the spontaneous breathing trial and at the end of the spontaneous breathing trial in critically ill patients undergoing mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Mechanical ventilation weaning success | 48 hours
  Weaning success: stable without mechanical ventilator support during more than 48 hours
Mechanical ventilation weaning failure | 48 hours
  Weaning failure: unstable without mechanical ventilator support within 48 hours

SECONDARY OUTCOMES:
Mortality | ICU mortality after ultrasonography guided weaning
  Incidence of ICU mortality

CONTACTS AND LOCATIONS:
Overall Officials: Şule Asrı, Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)

REFERENCES:
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Background] Dres M, Goligher EC, Heunks LMA, Brochard LJ. Critical illness-associated diaphragm weakness. Intensive Care Med. 2017 Oct;43(10):1441-1452. doi: 10.1007/s00134-017-4928-4. Epub 2017 Sep 15. PMID 28917004